CLINICAL TRIAL: NCT06806826
Title: Evaluatıon of the Effectıveness of Omalızumab Treatment In Patıents Wıth Allergıc Rhınıtıs
Brief Title: The Effect of Omalizumab on Allergic Rhinitis Symptoms: a Comparative Study
Acronym: rhinitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Semra Ağırbaş, asst.prof.dr, Yuzuncu Yil University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19.12.2018/09
Record Dates: First submitted 2025-01-21; First posted 2025-02-04 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Allergic Rhinitis
Keywords: allergic rhinitis; omalizumab
MeSH Terms: conditions — Rhinitis, Allergic | interventions — Omalizumab; montelukast

STUDY DESIGN:
Intervention Model Description: Between December 2018 and November 2019, 25 patients with both allergic rhinitis and chronic urticaria and 25 patients with allergic rhinitis only were included in the study. Patients with both allergic rhinitis and chronic urticaria received Omalizumab (300 mg/month) (Omalizumab group), while patients with allergic rhinitis received Montelukast 10 mg plus Desloratadine 5 mg daily (Desloratadine group). In addition, both groups received fluticasone propionate nasal spray (100 mcg/day in each nostril). At baseline and 8-10 weeks after the start of treatments (follow-up), allergic rhinitis symptoms such as nasal congestion, rhinorrhea, sneezing, and itchy eyes and quality of life were assessed. A self-report measure, a 10-cm linear visual analog scale (VAS), was used for the assessments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Omalizumab group (Active Comparator): Between December 2018 and November 2019, 25 patients with allergic rhinitis and chronic urticaria and 25 patients with allergic rhinitis only were included in the study. Patients with allergic rhinitis and chronic urticaria received Omalizumab (300 mg/month) (Omalizumab group).
  Interventions: Drug: Omalizumab
- (Desloratadine group). (Active Comparator): patients with allergic rhinitis received Montelukast 10 mg plus Desloratadine 5 mg daily (Desloratadine group).
  Interventions: Drug: Omalizumab

INTERVENTIONS:
Drug: Omalizumab — The patients in the study group were started on omalizumab and intranasal fluticasone propionate. Omalizumab was administered subcutaneously to these patients at a dose of 300 mg once a month. . Twenty-five patients in the control group were started on intranasal fluticasone propionate spray and a tablet containing 5 mg desloratadine+10 mg montelukast sodium at the same dose and in the same manner as the patients in the study group. The patients were asked to use 100 mg of suspension equivalent to 50 micrograms of fluticasone propionate as two sprays into each nostril once daily and to use the tablet once daily. Patients in both groups were asked to fill out the visual analog scale and their total Ig E levels were checked. Patients who were called for a check-up after eight to ten weeks were evaluated again with the visual analog scale.
  Other Names: desloratadin + montelukast

SUMMARY:
We aimed to evaluate the usability and efficacy of omalizumab in allergic rhinitis and its potential as an alternative treatment option.

DETAILED DESCRIPTION:
The study was conducted to determine the effectiveness of omalizumab on symptoms in patients diagnosed with allergic rhinitis and to compare it with current medical treatment options.

ELIGIBILITY:
Inclusion Criteria:

* Those who gave informed consent and wanted to participate in the study and did not have any additional systemic or nasal diseases were included.

Exclusion Criteria:

* under 18 years old,
* over 65 years old,
* with systemic comorbidities (diabetes mellitus, hypertension, chronic renal failure, hypothyroidism, etc.)
* patients with rhinosinusitis, nasal polyps, nasal septal deviation, tumors, smoking and nasal surgery, and non-compliant patients were excluded from this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
omalizumab treatment process | Patients were followed up for 3 months after starting treatment.
  Vas scores including runny nose, nasal congestion, sneezing, tearing and itching in the eyes were compared before and 3 months after omalizumab treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Yuzuncu Yıl üniversity dursun odabaş medical center, Van, tuşba, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No